CLINICAL TRIAL: NCT02232074
Title: Project SUPPORT (Socio-legal Services for Underserved Populations Through Patient Navigation to Optimize Resources During Treatment)
Brief Title: Socio-legal Services for Underserved Populations Through Patient Navigation to Optimize Resources During Treatment
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Battaglia, Tracy, Associate Professor of Medicine and Epidemiology, Boston University School of Medicine, Chief of Women's Health Unit, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-32599; RSG-13-368-01-CPPB (Other Grant/Funding Number: American Cancer Society); AD-1304-6272 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: Patient Navigation; Medical Legal Partnership; Healthcare Disparities
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient navigation enhanced with legal support (Experimental): In addition to receiving standard navigation, patients will be connected with a Patient Navigator who is partnered with a lawyer from Medical-Legal Partnership to provide personalized assistance with regard to social-legal barriers.
  Interventions: Other: Patient navigation enhanced with legal support
- Standard patient navigation (No Intervention): These patients will receive standard patient navigation which will work to ensure that services are coordinated amongst medical personnel, while also addressing patients' needs.

INTERVENTIONS:
Other: Patient navigation enhanced with legal support
  Arms: Patient navigation enhanced with legal support

SUMMARY:
The investigators plan to compare standard patient navigation with an enhanced navigation partnered with the Medical Legal Partnership | Boston (MLP) to determine if assessing legal needs of newly diagnosed cancer patients in addition to other barriers to care leads to better clinical outcomes.

DETAILED DESCRIPTION:
Differences and delays in the delivery of cancer care lead to more advanced cancer at the time of diagnosis and ultimately to more deaths for low-income and minority communities. Our group helped develop a patient-navigation model using lay health workers to address patient barriers and coordinated cancer-care services, leading to more timely care. Despite the fact that patient navigation is now a standard required by the Commission on Cancer, the investigators' research shows that delays in care persist for our low-income patients with socio-legal barriers. Socio-legal barriers are defined as social problems related to meeting life's most basic needs that are supported by public policy or programming and thus potentially remedied through legal advocacy/action (e.g., unsafe/unstable housing, unlawful utility shutoffs, or job termination). Direct feedback from cancer patients suggests a critical need to address socio-legal barriers in order to achieve quality care for all. To expand the current impact of patient navigation on quality care for low-income patients, the investigators will partner with patients, key community stakeholders, and the Medical-Legal Partnership (MLP)|Boston, the founding site of a nationwide program assisting healthcare teams in addressing socio-legal barriers to health. Under direction from a Patient Advisory Group and a Community Advisory Board, the investigators will conduct a study to compare standard navigation with an MLP navigation intervention enhanced by legal support for low-income cancer patients.

The investigators will enroll 374 low-income, racially diverse, newly diagnosed cancer patients. Half will receive standard navigation, i.e., a lay navigator integrated into the healthcare team who provides one-on-one patient contact to address traditional system barriers to care. The other half will receive MLP navigation, i.e., standard navigation enhanced by legal support including:

1. a full socio-legal needs assessment and care plan in consultation with MLP; and
2. legal assistance for eligible urgent legal needs. We will compare each group on all outcomes.

Compared to standard navigation, we expect that addressing socio-legal barriers to care with MLP navigation will improve patient-reported outcomes and lead to more timely care delivery. Because of widespread national availability of patient navigation and MLP programs at hospitals serving vulnerable patients, this intervention can be quickly replicated to improve patient experience and survival.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast and lung cancer patients
* Within 30 days of patient being informed of diagnosis
* Receiving cancer care at Boston Medical Center
* No history of cancer treatment in past 5 years
* No cognitive impairments
* Over 18 years of age
* Speak English, Spanish or Haitian Creole

Exclusion Criteria:

* Patient informed of cancer diagnosis >30 days
* Patient under 18 yrs. of age
* Primary language something other than English, Spanish or Haitian Creole
* Undergoing treatment for concurrent cancer
* Patient has history of cancer or has received cancer treatment within the last 5 years
* Institutionalized/cognitive impairment (such as: dementia or metabolic, medication or drug induced), given the unique challenges to their treatment decision making/adherence and the fact that the intervention would not include the patient directly, but rather the family.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Battaglia, M.D., M.P.H, Principal Investigator — Boston Medical Center; Sharon Bak, M.P.H, Study Director — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Navigation With Legal Support: For those with legal concerns at baseline identified by the IHELP screening tool, intervention participants received Patient Navigation enhance with legal support.
- Standard Patient Navigation: For those with legal concerns at baseline identified by the IHELP screening tool, control participants received standard of care Patient Navigation
Period: Overall Study
Arm/Group | Patient Navigation With Legal Support | Standard Patient Navigation
Started | 154 | 152
Completed | 113 | 107
Not Completed | 41 | 45
Not completed — Withdrawal by Subject | 5 | 3
Not completed — No legal concerns at baseline | 36 | 41
Not completed — deemed ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis includes those participants with at least 1 legal concern at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Navigation With Legal Support | Standard Patient Navigation | Total
Number analyzed (Participants) | 113 | 107 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis includes those participants with at least 1 legal concern at baseline.
  years | 55.6 (11.0) | 54.7 (11.0) | 55.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 102 | 211
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White | 26 | 27 | 53
  Race / Ethnicity: Hispanic | 22 | 26 | 48
  Race / Ethnicity: Black \ African-American | 60 | 51 | 111
  Race / Ethnicity: Other | 5 | 3 | 8
Language [Count of Participants; unit: Participants]
  English | 87 | 71 | 158
  Spanish | 17 | 27 | 44
  Haitian Creole | 9 | 9 | 18
Insurance [Count of Participants; unit: Participants]
  Public | 83 | 79 | 162
  Private | 30 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Initiating Treatment Within 90 Days of Diagnosis Among BREAST Cancer Participants
Description: The receipt of timely care will be defined as initiation of care within 90 days, as this the shortest delay that has been shown to consistently affect mortality The time element was calculated from date of diagnosis (Time0) to date of treatment initiation (Time1) .The date chosen for the Time1 variable depends on the recommended care plan for each patient, as derived from the chart abstraction and based on patient presentation.
Time Frame: Receipt of 1st treatment within 90 days from diagnosis
Population: breast cancer participants with 1 or more legal concern as screened at baseline using the IHELP survey.
Measure: Count of Participants; unit: Participants
Groups:
- Breast Cancer Intervention: For breast cancer participants with at least 1 legal concern at baseline, intervention participants received patient navigation enhanced with legal support.
- Breast Cancer Control: For breast cancer participants with at least 1 legal concern at baseline, control participants received standard of care patient navigation.
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 98 | 96
Participants | 94 | 92
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Compared to the control group, the Breast cancer INTERVENTION group will be more likely to have timely first treatment (i.e. receipt of first treatment within 90 days of diagnosis); Test type: Superiority; p = 0.77, Regression, Logistic — a priori threshold for statistical significance p<0.05; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.21 to 3.14]

2. Primary Outcome: Proportion of Participants Initiating Treatment Within 90 Days of Diagnosis Among LUNG Cancer Participants
Description: as for outcome 1
Time Frame: Receipt of 1st treatment within 90 days from diagnosis
Measure: Count of Participants; unit: Participants
Groups:
- Lung Cancer Intervention: For lung cancer participants with at least 1 legal concern at baseline, intervention participants received patient navigation enhanced with legal support.
- Lung Cancer Control: For lung cancer participants with at least 1 legal concern at baseline, control participants received standard of care patient navigation.
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 8 | 11
Participants | 7 | 7
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Compared to the control group, the Lung cancer INTERVENTION group will be more likely to have timely first treatment (i.e. receipt of first treatment within 90 days of diagnosis); Test type: Superiority; p = 0.26, Regression, Logistic — a priori threshold for statistical significance p<0.05; Odds Ratio (OR) = 4.00, 95% CI 2-sided [0.35 to 45.4]

3. Secondary Outcome: Distress Thermometer at 3 Months for BREAST Cancer Patients
Description: Distress will be assessed through patient interviews utilizing the Distress Thermometer (DT) instrument with a scale from 0 (no distress) to 10 (extreme distress). Lower values are more favorable.
Time Frame: 3 months after enrollment
Population: The number of Intervention participants decreased by 5 to 99 and Control participants decreased by 3 to 90 due to missing Distress Thermometer data at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 99 | 90
units on a scale | 5.60 (3.20) | 5.90 (3.00)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Compared to the control group, the Breast cancer INTERVENTION group will have less distress at 3 months post-enrollment; Test type: Superiority; p = 0.53, Regression, Linear — a priori threshold for statistical significance p<0.05; Adjusting for baseline Distress Thermometer scores; Median Difference (Final Values) = -0.27, Standard Error of Mean 0.42

4. Secondary Outcome: Distress Thermometer at 3 Months for LUNG Cancer Patients
Description: as for outcome 3
Time Frame: 3 months after enrollment
Population: The number of LUNG Control participants decreased by 3 for a total of 8 due to missing Distress Thermometer data at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 8 | 8
units on a scale | 4.50 (3.20) | 6.10 (2.70)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Compared to the control group, the LUNG cancer INTERVENTION group will have less distress at 3 months post-enrollment; Test type: Superiority; p = 0.43, Regression, Linear — Adjusting for baseline Distress Thermometer scores; Median Difference (Final Values) = -1.32, Standard Error of Mean 1.62

5. Secondary Outcome: Distress Thermometer at 6 Months for BREAST Cancer Patients
Description: as for outcome 3
Time Frame: 6 months after enrollment
Population: The number of BREAST Intervention participants decreased by 13 for a total of 91 and Control participants decreased by 8 for a total of 58 due to missing Distress Thermometer data at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 91 | 85
units on a scale | 4.50 (3.30) | 5.20 (3.00)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Compared to the control group, the Breast cancer INTERVENTION group will have less distress at 6 months post-enrollment; Test type: Superiority; p = 0.18, Regression, Linear — a priori threshold for statistical significance p<0.05; Adjusting for baseline Distress Thermometer scores; Median Difference (Final Values) = -0.60, Standard Error of Mean 0.45

6. Secondary Outcome: Distress Thermometer at 6 Months for LUNG Cancer Patients
Description: Distress will be assessed through patient interviews utilizing the Distress Thermometer (DT) instrument with a scale from 0 (no distress) to 10 (extreme distress).Lower values are more favorable.
Time Frame: 6 months after enrollment
Population: The number of LUNG Intervention participants decreased by 2 for a total of 6 and Control patients decreased by 4 due to missing Distress Thermometer data at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 6 | 7
units on a scale | 1.50 (1.90) | 4.00 (2.60)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Compared to the control group, the Lung cancer INTERVENTION group will have less distress at 6 months post-enrollment; Test type: Superiority; p = 0.33, Regression, Linear — a priori threshold for statistical significance p<0.05; Adjusting for baseline Distress Thermometer scores; Median Difference (Final Values) = -1.33, Standard Error of Mean 1.29

7. Secondary Outcome: Cancer Needs and Distress Inventory at 6 Months for BREAST Cancer Patients
Description: Patient needs were assessed through patient interviews utilizing the Cancer Needs Distress Inventory (CaNDI) instrument. The CaNDI is a 38-item self-report instrument that rates need and distress level in the past two weeks using a 5 -point Likert scale where 1=not a problem to 5=very severe problem. For this analysis, the mean total score is reported with the minimum value=1 and the maximum value=4.10. Lower values are more favorable.
Time Frame: 6 months post-enrollment
Population: The number of Breast Intervention participants decreased by 13 to 91 and the Control participants decreased by 8 to 85 due to missing CaNDi data at 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 91 | 85
score on a scale | 1.70 (0.70) | 1.70 (0.60)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Test type: Superiority; p = 0.68, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = 0.03, Standard Error of Mean 0.07

8. Secondary Outcome: Cancer Needs and Distress Inventory at 6 Months for LUNG Cancer Patients
Description: Patient needs were assessed through patient interviews utilizing the Cancer Needs Distress Inventory (CaNDI) instrument. The CaNDI is a 38-item self-report instrument that rates need and distress level in the past two weeks using a 5 -point Likert scale where 1=not a problem to 5=very severe problem. For this analysis, the mean total score is reported with the minimum value=1 and the maximum value=2.3. Lower values are more favorable.
Time Frame: 6 months post-enrollment
Population: The number of Lung Intervention participants decreased by 2 to 6 and the Control participants decreased by 4 to 7 due to missing CaNDi data at 6 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 6 | 7
score on a scale | 1.40 (0.40) | 1.50 (0.50)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Test type: Superiority; p = 0.26, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = -0.18, Standard Error of Mean 0.15

9. Secondary Outcome: Patient Satisfaction With Navigation at 6 Months Among BREAST Cancer Patients
Description: Patient's satisfaction assessed through the Patient Satisfaction with Interpersonal Relationship with Navigator Measure (PSN-1) questionnaire. Each question of the 9-item instrument has a 5 point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Responses are summed for a total score. The higher the score, the higher patient's satisfaction with navigation. The minimum value=9 and the maximum value=45. Higher values are more favorable.
Time Frame: 6 months post-enrollment
Population: Linear regression tested for an association between the intervention & control groups in satisfaction with patient navigation at six months post-enrollment. The number of Breast Intervention participants decreased by 52 to 52 and the Control participants decreased by 41 to 52 due to missing Patient Satisfaction data at 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 52 | 52
units on a scale | 40.4 (7.44) | 39.7 (7.00)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Compared to the control group, the Breast cancer INTERVENTION group will be more satisfied with patient navigation at 6 months post-enrollment; Test type: Superiority; p = 0.62, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = 0.71, Standard Error of Mean 1.43

10. Secondary Outcome: Patient Satisfaction With Navigation at 6 Months Among LUNG Cancer Patients
Description: as for outcome 9
Time Frame: 6 months post-enrollment
Population: Linear regression tested for an association between the intervention & control groups in satisfaction with patient navigation at six months post-enrollment. The number of LUNG Intervention participants decreased by 4 to 4 and the Control participants decreased by 8 to 3 due to missing Patient Satisfaction data at 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 4 | 3
units on a scale | 40.3 (4.43) | 39.0 (2.65)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Compared to the control group, the Lung cancer INTERVENTION group will be more satisfied with patient navigation at 6 months post-enrollment; Test type: Superiority; p = 0.69, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = 1.25, Standard Error of Mean 2.91

11. Secondary Outcome: Self-efficacy for BREAST Cancer Patients at 6 Months
Description: Self-Efficacy will be assessed through patient interviews utilizing the Communication and Attitudinal Self-Efficacy (CASE). The CASE is a 12-item instrument that rates self-efficacy in three domains: (1) seeking and obtaining information, (2) understanding and participating in care, and (3) maintaining a positive attitude. Total scores range from 12 to 48. A higher score is more favorable, indicating a positive attitude and strong self-efficacy.
Time Frame: 6 months post-enrollment
Population: Within each cancer group (breast & lung cancers analyzed separately), a linear regression was used to test whether there was an association between the intervention & control groups in self-efficacy at six months post-enrollment, adjusting for baseline CASE Cancer score.
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 90 | 83
total score on a scale | 44.0 (5.2) | 43.3 (4.9)
Statistical Analysis 1: Comparison: Breast Cancer Intervention; Compared to the control group, the breast cancer INTERVENTION group would have higher self-efficacy was adjusting for baseline self-efficacy scores; Test type: Superiority; p = 0.58, Regression, Linear — a priori threshold for statistical significance p<0.05; adjusting for baseline Case scores; Median Difference (Final Values) = 0.33, Standard Error of Mean 0.59

12. Secondary Outcome: Self-efficacy for LUNG Cancer Patients at 6 Months
Description: as for outcome 11
Time Frame: 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 6 | 7
total score on a scale | 47.0 (0.90) | 43.0 (5.00)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Compared to the control group, the lung cancer INTERVENTION group would have higher self-efficacy was adjusting for baseline self-efficacy scores; Test type: Superiority; p = 0.09, Regression, Linear; adjusting for baseline Case scores; Median Difference (Final Values) = 4.20, Standard Error of Mean 2.21

13. Secondary Outcome: Number of Participants Receiving Radiation Within 365 Days of Cancer Diagnosis
Description: The receipt of quality care is defined as receiving radiation to the breast within one year of a breast cancer diagnosis if: under the age of 70, estrogen or progesterone tumor positive and had breast conserving surgery.
Time Frame: Measured at 12 months
Population: Excluded those women who did not meet requirements for receipt of radiation: over 70 years of age, with tumor negative for estrogen or progesterone
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 57 | 66
Participants | 6 | 6
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; We hypothesize that compared to the control group, the Breast cancer INTERVENTION group will receive quality care (i.e. receipt of radiation within one year of diagnosis); Test type: Superiority; p = 0.79, Regression, Logistic — a priori threshold for statistical significance p<0.05; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.28 to 2.79]

14. Secondary Outcome: Distress Thermometer at 12 Months for BREAST Cancer Patients
Description: as for outcome 3
Time Frame: 12 months after enrollment
Population: The number of BREAST Intervention participants decreased by 22 for a total of 82 and Control participants decreased by 18 for a total of 75 due to missing Distress Thermometer data at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 82 | 75
units on a scale | 5.3 (3.5) | 5.3 (3.3)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; We hypothesize that compared to the control group, the Breast cancer INTERVENTION group will have less distress at 12 months post-enrollment; Test type: Superiority; p = 0.71, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = 0.19, Standard Error of Mean 0.50

15. Secondary Outcome: Distress Thermometer at 12 Months for LUNG Cancer Patients
Description: Distress will be assessed through patient interviews utilizing the Distress Thermometer (DT) instrument with a scale from 0 (no distress) to 10 (extreme distress). Lower scores are more favorable.
Time Frame: 12 months after enrollment
Population: The number of LUNG Intervention participants decreased by 3 for a total of 5. Control participants decreased by 6 for a total of 5 due to missing data at 12 months follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 5 | 5
units on a scale | 3.6 (3.0) | 6.0 (4.7)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; We hypothesize that compared to the control group, the Lung cancer INTERVENTION group will have less distress at 12 months post-enrollment; Test type: Superiority; p = 0.61, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = -1.45, Standard Deviation 2.71

16. Secondary Outcome: Cancer Needs and Distress Inventory at 12 Months for BREAST Cancer Patients
Description: Patient needs were assessed through patient interviews utilizing the Cancer Needs Distress Inventory (CaNDI) instrument. The CaNDI is a 38-item self-report instrument that rates need and distress level in the past two weeks using a 5 -point Likert scale where 1=not a problem to 5=very severe problem. The mean total score is reported.
Time Frame: 12 months post-enrollment
Population: The number of BREAST Intervention participants decreased by 23 for a total of 81. The Control participants decreased by 18 for a total of 75 due to missing CaNDI data at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 81 | 75
score on a scale | 1.70 (0.70) | 1.70 (0.60)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Test type: Superiority; p = 0.46, Regression, Linear — a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = 0.06, Standard Deviation 0.08

17. Secondary Outcome: Cancer Needs and Distress Inventory at 12 Months for LUNG Cancer Patients
Description: as for outcome 16
Time Frame: 12 months post-enrollment
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lung Cancer Intervention: Lung cancer participants with at least 1 legal concern at baseline, intervention participants received patient navigation enhanced with legal support.
- Lung Cancer Control: Lung cancer participants with at least 1 legal concern at baseline, control participants received standard of care patient navigation.
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 5 | 5
score on a scale | 1.50 (0.70) | 1.50 (0.40)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Test type: Superiority; p = 0.89, Regression, Linear — a priori threshold for statistical significance p<0.05; Median Difference (Final Values) = -0.03, Standard Deviation 0.20

18. Secondary Outcome: Patient Satisfaction With Navigation at 12 Months Among BREAST Cancer Patients
Description: Patient's satisfaction assessed through the Patient Satisfaction with Interpersonal Relationship with Navigator Measure (PSN-1) questionnaire. Each question of the 9-item instrument has a 5 point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Responses are summed for a total score. The higher the score, the higher patient's satisfaction with navigation. The minimum value=9 and the maximum value=45. Higher scores are more favorable.
Time Frame: 12 months post-enrollment
Population: The number of BREAST Intervention participants decreased by 52 for a total of 52 and Control participants decreased by 55 for a total of 38 due to missing data at 12 months post-enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 52 | 38
score on a scale | 40.8 (6.9) | 38.4 (8.9)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Test type: Superiority; p = 0.16, Regression, Linear — a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = 2.38, Standard Deviation 1.66

19. Secondary Outcome: Patient Satisfaction With Navigation at 12 Months Among LUNG Cancer Patients
Description: as for outcome 18
Time Frame: 12 months post-enrollment
Population: The number of Lung Intervention participants decrease by 5 for a total of 3 and the number of Lung Control participants decreased by 7 for a total of 4 due to missing data at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 3 | 4
score on a scale | 37.7 (2.9) | 42.5 (4.4)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Test type: Superiority; p = 0.16, Regression, Linear — a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = -4.83, Standard Deviation 2.93

20. Secondary Outcome: Self-efficacy for BREAST Cancer Patients at 12 Months
Description: Self-Efficacy will be assessed through patient interviews utilizing the Communication and Attitudinal Self-Efficacy (CASE). The CASE is a 12-item instrument that rates self-efficacy in three domains: (1) seeking and obtaining information, (2) understanding and participating in care, and (3) maintaining a positive attitude. A higher score indicates a positive attitude and strong self-efficacy. Total scores range from 12 to 48. A higher score is more favorable, indicating a positive attitude and strong self-efficacy.
Time Frame: 12 months post-enrollment
Population: The number of BREAST Intervention participants decreased by 23 for a total of 81 and for control participants by 19 for a total of 74 due to missing values at 12 months post-enrollment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Breast Cancer Intervention | Breast Cancer Control
Number analyzed (Participants) | 81 | 74
score on a scale | 44.2 (4.5) | 43.0 (5.6)
Statistical Analysis 1: Comparison: Breast Cancer Intervention vs Breast Cancer Control; Test type: Superiority; p = 0.13, Regression, Linear — a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = 1.14, Standard Deviation 0.75

21. Secondary Outcome: Self-efficacy for LUNG Cancer Patients at 12 Months
Description: as for outcome 20
Time Frame: 12 months post-enrollment
Population: The number of Lung Intervention participants decrease by 3 for a total of 5 and the number of Lung Control participants decreased by 6 for a total of 5 due to missing data at 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lung Cancer Intervention | Lung Cancer Control
Number analyzed (Participants) | 5 | 5
score on a scale | 44.2 (4.8) | 43.6 (5.5)
Statistical Analysis 1: Comparison: Lung Cancer Intervention vs Lung Cancer Control; Test type: Superiority; p = 0.80, Regression, Linear — a priori threshold for statistical significance p<0.05; Mean Difference (Final Values) = 0.97, Standard Deviation 3.70

ADVERSE EVENTS:
Time Frame: Study enrollment began 2/1/2014 and ended 9/30/2018. Participants were assessed throughout their study participation to 1 year after enrollment.
Description: Involvement in this study has minimal risks. The main potential risk of this study is loss of confidentiality. As multiple safeguards were in place, including keeping files in a locked cabinets and only conducting data analysis on a data set that is coded and does not contain any direct identifiers.
Arm/Group | Patient Navigation With Legal Support | Standard Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/107
Other Adverse Events (participants affected / at risk) | 0/113 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT02232074/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02232074/Prot_ICF_001.pdf